CLINICAL TRIAL: NCT04393012
Title: Voxello - V-1, Alternative Nurse Call
Brief Title: Providing Access to an Alternative Nurse Call
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa Adaptive Technologies, Inc. (Industry)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Voxello V1; R44NR016406 (NIH)
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Problems With Access to Health Care
Keywords: alternative access; patient-provider communication

STUDY DESIGN:
Intervention Model Description: Evaluation of impact
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Noddle Group (Experimental): Patients who received noddle to allow access to the nurse call system.
  Interventions: Other: Provide alternative nurse call and communication device

INTERVENTIONS:
Other: Provide alternative nurse call and communication device — Evaluate impact of providing access to the nurse call system and a speech generating device.

SUMMARY:
To address the needs of the many patients who cannot access the standard nurse call systems Iowa Adaptive Technologies has developed the Noddle, a smart switch that can take the smallest intentional gesture a patient can make (e.g. tongue click, wink) and allow the patient to access the nurse call system and control a speech-generating device. This study will assess how patients and their nurses as well as family members perceive the impact of having a device that would allow them to summon the nurse and to be able to effectively communicate. Patients will be provided a Noddle and will be free to use it as much or a little as they like during their hospitalization. Patients will either use the Noddle just to access the nurse call system or they will use it to access the nurse call system and a speech-generating device. Patients, nurses and family members will be asked to complete an exit questionnaire prior to discharge from the hospital.

DETAILED DESCRIPTION:
The study will evaluate the responses of patients, nurses and family members to the use of the Noddle switch to enable the patients to access the nurse call system and a speech generating device. Patients who cannot access the standard nurse call and who may not be able to speak due to mechanical ventilation will be recruited to the study and provided the opportunity to use the Noddle switch as long as they want while they are hospitalized at UIHC. Prior to their discharge or when they no longer need or want to use the Noddle switch, they along with their nurses and family members (if present) will be asked to complete a survey to assess their ability to effectively communicate. The data from the study participants will be compared to data from two groups of patients from a previous study who were either able to or unable to access the nurse call system and communicate with caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be conscious, able to produce an intentional gesture and appropriately respond to yes/no questions.
2. Patients must be severely limited in their mobility and unable to access the nurse call system and/or must be unable to use normal modes of oral and written modes of communication.

Exclusion Criteria:

1. Patients who are sedated or unconscious (patients who are sedated for limited time may be considered).
2. Can access the nurse call and speak without other assistance

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Exit Survey Responses | Completed on the 1 day the patient finished use of the device(s).
  Patient and Nurse Exit Surveys

CONTACTS AND LOCATIONS:
Overall Officials: Richard R Hurtig, Ph.D., Principal Investigator — Iowa Adaptive Technologies Inc. (dba Voxello)

IPD SHARING:
Plan to Share IPD: No
De-identified survey results are stored and could be shared as Excel files